CLINICAL TRIAL: NCT04189588
Title: A Phase 2 Exploratory Study of Intravenous QUZYTTIR™ (Cetirizine Hydrochloride Injection) Versus Intravenous Diphenhydramine in the Prevention of Hypersensitivity Infusion Reactions
Brief Title: Phase 2 Study IV QUZYTTIR™ (Cetirizine Hydrochloride Injection) vs V Diphenhydramine
Acronym: versus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TerSera Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TER-QZTR-001
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Oncology Patients Receiving Chemotherapy
MeSH Terms: interventions — Cetirizine; Diphenhydramine; Rituximab; Paclitaxel; ofatumumab; ocrelizumab; obinutuzumab; ibritumomab tiuxetan

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Active Comparator): Cetirizine HCl 10 mg/mL: a single 1 mL injection.
  Interventions: Drug: Cetirizine HCl 10 mg/mL; Drug: anti-CD20 such as Rituximab or Paclitaxel
- Cohort B (Active Comparator): Diphenhydramine 50 mg/mL: a single 1 mL injection.
  Interventions: Drug: Diphenhydramine 50 mg/mL; Drug: anti-CD20 such as Rituximab or Paclitaxel

INTERVENTIONS:
Drug: Cetirizine HCl 10 mg/mL — Comparison of two injectable products: cetirizine HCl 10 mg/mL and diphenhydramine 50 mg/mL, both administered during a 1 to 2-minute period by IV push using a 1 mL syringe
  Other Names: Quzyttir™
  Arms: Cohort A
Drug: Diphenhydramine 50 mg/mL — Comparison of two injectable products: cetirizine HCl 10 mg/mL and diphenhydramine 50 mg/mL, both administered during a 1 to 2-minute period by IV push using a 1 mL syringe
  Other Names: Benadryl injection®
  Arms: Cohort B
Drug: anti-CD20 such as Rituximab or Paclitaxel — Compare the number of infusion reactions to treatment with an anti-CD20 such as Rituxan® (Rituximab) or Taxol® (Paclitaxel) after premedication with intravenous (IV) QUZYTTIR™ cetirizine hydrochloride (HCl) or IV diphenhydramine during first-cycle infusion or re-treatment. Re-treatment is defined as re-treatment with Rituxan® (Rituximab) or Paclitaxel after 6 months in patients with persistent infusion reactions while on maintenance or re-treatment.
  Other Names: Rituxan®; Taxol; Arzerra; Ocrevus; Gazyva; Ruxience; Truxima; Zevalin

SUMMARY:
This study is designed to compare the number of infusion reactions to treatment with an anti-CD20 such as Rituxan® (rituximab) or Taxol® (Paclitaxel) after premedication with intravenous (IV) QUZYTTIR™ cetirizine hydrochloride (HCl) or IV diphenhydramine during first-cycle infusion or re-treatment with an anti-CD20 such as Rituxan® (rituximab) or Paclitaxel. Re-treatment is defined as re-treatment with an anti-CD20 such as Rituxan® (rituximab) or Paclitaxel after 6 months or in patients with persistent infusion reactions while on maintenance or retreatment.

DETAILED DESCRIPTION:
This will be a randomized, double-blind exploratory study of IV cetirizine HCl 10 mg/mL versus IV diphenhydramine 50 mg/mL in approximately 34 patients who require premedication for hypersensitivity infusion reactions associated with an anti-CD20 such as Rituxan® (rituximab) or Paclitaxel. The objectives and purpose of the study will be described to patients presenting at the participating infusion centers. The patients will be randomized to receive either IV cetirizine HCl or IV diphenhydramine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who require treatment premedication with an antihistamine for hypersensitivity infusion reactions associated with an anti-CD20, such as Rituxan® (Rituximab) or Paclitaxel, in their first-cycle or re-treatment after 6 months or in patients with persistent infusion reactions while on maintenance or re-treatment.
* 18 years of age or older

Exclusion Criteria:

* Receipt of an investigational drug or device within the past 30 days.
* Patients with likelihood of developing or history of tumor lysis syndrome.(TLS): patients with auto-lyse, Burkitt lymphoma and diffuse large B-cell lymphoma (DLBCL) with bulky disease (single node 7 or more cm or 3 or more nodal sites with size 3 or more cm)
* Patients in whom an antihistamine may be contraindicated (e.g., narrow angle glaucoma, symptomatic prostatic hypertrophy).
* Patients who, in the opinion of the investigator, may not tolerate an IV injection of diphenhydramine 50 mg or cetirizine HCl 10 mg.
* Receipt of any antihistamine (H1 antagonist) within the past 2 hours regardless of the route of administration, e.g., diphenhydramine, cetirizine, loratadine, fexofenadine, levocetirizine, desloratadine. chlorpheniramine, clemastine, and doxylamine
* Receipt of an H2 antagonist within the past 4 hours, e.g., ranitidine, cimetidine, famotidine, nizatidine.
* Receipt of doxepin within the past 24 hours; doxepin is an antidepressant, but it also has antihistamine properties.
* Receipt of epinephrine (EpiPen® or any other brand) within the past 30 days.
* Has known allergy to hydroxyzine, cetirizine, or levocetirizine, or diphenhydramine.
* Pregnant or breastfeeding.
* Any condition that in the view of the investigator makes the patient unsuitable for enrollment in this study.
* Major medical or psychiatric illness, other than diagnosed cancer at the time of presentation or in the past that in the investigator's judgement they should not be enrolled in this clinical trial.
* Inability to provide informed consent.
* Patients on concomitant P-glycoprotein inhibitors; including antidepressants, antipsychotics (e.g., olanzapine), and benzodiazepines (e.g., alprazolam), as they may cause an increase in sedation.
* Receipt of drugs that cause sedation within the past 24 hours prior to administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janine North, B.S., Study Director — TerSera Therapeutics
Locations (7):
- United States (7):
  - St.Joseph Heritage Care, Napa, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Oncology Consultants, Houston, Texas
  - Baylor, Scott, & White Medical Center, Round Rock, Texas
  - Baylor, Scott, & White Medical Center, Temple, Texas
  - Baylor, Scott, & White Medical Center, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmes JP, Peguero JA, Garland RC, North J, Young S, Brent LD, Joseph-Ridge N. Intravenous Cetirizine vs Intravenous Diphenhydramine for the Prevention of Hypersensitivity Infusion Reactions: Results of an Exploratory Phase 2 Study. J Infus Nurs. 2021 Nov-Dec 01;44(6):315-322. doi: 10.1097/NAN.0000000000000444. PMID 34555839
- See also: Results Publication in Journal of Infusion Nursing: Intravenous Cetirizine vs Intravenous Diphenhydramine for the Prevention of Hypersensitivity Infusion Reactions: Results of an Exploratory Phase 2 Study — https://journals.lww.com/journalofinfusionnursing/Fulltext/2021/11000/Intravenous_Cetirizine_vs_Intravenous.2.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Cetirizine HCl 10 mg/mL: a single 1 mL injection.
  Diphenhydramine 50 mg/mL: Comparison of two injectable products: cetirizine HCl 10 mg/mL and diphenhydramine 50 mg/mL, both administered during a 1 to 2-minute period by IV push using a 1 mL syringe
  anti-CD20 such as Rituximab or Paclitaxel: Compare the incidence of infusion reactions to treatment with an anti-CD20 such as Rituxan® (Rituximab) or Taxol® (Paclitaxel) after premedication with intravenous (IV) QUZYTTIR™ cetirizine hydrochloride (HCl) or IV diphenhydramine during first-cycle infusion or re-treatment. Re-treatment is defined as re-treatment with Rituxan® (Rituximab) or Paclitaxel after 6 months in patients with persistent infusion reactions while on maintenance or re-treatment.
- Cohort B: Diphenhydramine 50 mg/mL: a single 1 mL injection.
  Cetirizine HCl 10 mg/mL: Comparison of two injectable products: cetirizine HCl 10 mg/mL and diphenhydramine 50 mg/mL, both administered during a 1 to 2-minute period by IV push using a 1 mL syringe
  anti-CD20 such as Rituximab or Paclitaxel: Compare the incidence of infusion reactions to treatment with an anti-CD20 such as Rituxan® (Rituximab) or Taxol® (Paclitaxel) after premedication with intravenous (IV) QUZYTTIR™ cetirizine hydrochloride (HCl) or IV diphenhydramine during first-cycle infusion or re-treatment. Re-treatment is defined as re-treatment with Rituxan® (Rituximab) or Paclitaxel after 6 months in patients with persistent infusion reactions while on maintenance or re-treatment.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 17 | 17
Completed Treatment | 17 | 17
Completed (Completed 28-day Follow-up Period) | 17 | 15
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.83) | 66.6 (10.16) | 63.5 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Hypersensitivity Reactions to Treatment With an Anti-CD20 Antibody or Paclitaxel
Description: Compare the number of patients experiencing any infusion reaction events, and the number and percentage of patients experiencing each symptom of infusion reactions (ﬂushing, itching, alterations in heart rate and blood pressure, dyspnea, chest discomfort, acute back or abdominal pain, fever, shaking chills, nausea, vomiting, diarrhea, skin rashes, throat tightening, hypoxia, seizures, dizziness, or syncope) to treatment with anti-CD20 such as Rituxan® (rituximab) or Paclitaxel after premedication with intravenous (IV) QUZYTTIR™ cetirizine hydrochloride (HCl) or IV diphenhydramine during first-cycle infusion or re-treatment after 6 months or in patients with persistent infusion reactions while on maintenance with anti-CD20 such as Rituxan® (rituximab) or Paclitaxel.
  The infusion reactions will be evaluated following the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) deﬁnitions of graded infusion reactions.
Time Frame: During and after anti-CD20 agent or paclitaxel infusion, at 1 and 2 hours after the antihistamine injection, at time of discharge, and up through 1 Month post injection of antihistamine (intervention).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 17
Participants | 2 | 3

2. Secondary Outcome: Patient Sedation Scores at 1 Hour and 2 Hours Post-injection of Antihistamine (IV Cetirizine HCl or IV Diphenhydramine) and at Discharge.
Description: Patient sedation scores at 1 hour and 2 hours post-injection of antihistamine (IV cetirizine HCl or IV diphenhydramine) and at discharge. The patient sedation scores are assessed on a scale of 0-4, with 0=None and 4=Extremely Severe (Asleep, Cannot Self-Rate). The HCP sedation scores are assessed on a scale of 0-4, with 0=None and 4=Extremely severe.
Time Frame: 1 hour, 2 Hours and at discharge
Population: Per Patient Analysis set (patients with a baseline sedation score = 0)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 17
Units on a scale
  1 Hour | 0.5 (0.72) | 1.3 (1.26)
  2 Hour | 0.6 (0.61) | 0.9 (1.14)
  Discharge | 0.1 (0.33) | 0.4 (0.71)

3. Secondary Outcome: Time From Injection to "Readiness for Discharge"
Description: Describe the distribution of the amount of time spent in the treatment center prior to discharge (time from injection to "Readiness for Discharge").
Time Frame: Time to discharge from infusion center
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 17 | 17
Hours | 4.3 (1.54) | 4.7 (1.26)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=17) | Cohort B (N=17)
Septic Shock (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT04189588/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT04189588/SAP_001.pdf